CLINICAL TRIAL: NCT06968936
Title: Short-term Preoperative Combined Iron, Erythropoietin, and Vitamin C Therapy in Patients With Iron-deficiency Anaemia Undergoing Elective Cardiac Surgery: a Randomised Controlled Trial
Brief Title: Perioperative Blood Conservation: Role of Combined Iron Supplementation Protocols in Reducing Allogeneic Transfusion
Acronym: CIPAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20240384
Record Dates: First submitted 2025-04-13; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Anemia; Iron Deficiencies; Cardiac Surgery
MeSH Terms: conditions — Anemia; Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: Central stratified block group randomization
Who Masked: Outcomes Assessor
Masking Description: Blinding was maintained for outcome assessors, extracorporeal circulation staff, and all investigators not directly involved in the treatment process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Iron Supplementation Group (Experimental): Patients in the experimental group will receive a combination therapy consisting of intravenous sucrose iron (200 mg), subcutaneous recombinant human erythropoietin (150 IU/kg), and intravenous vitamin C (2 g), administered once daily for three consecutive days within the week prior to surgery. All perioperative transfusion decisions will follow standardized restrictive transfusion thresholds
  Interventions: Drug: Sucrose Iron，subcutaneous recombinant human erythropoietin，intravenous vitamin C
- Conventional treatment group (Active Comparator): Routine perioperative management based on clinical judgment, including observation, monitoring, and standard nursing practices
  Interventions: Procedure: Routine perioperative management

INTERVENTIONS:
Drug: Sucrose Iron，subcutaneous recombinant human erythropoietin，intravenous vitamin C — Patients in the experimental group will receive a combination therapy consisting of intravenous sucrose iron (200 mg), subcutaneous recombinant human erythropoietin (150 IU/kg), and intravenous vitamin C (2 g), administered once daily for three consecutive days within the week prior to surgery.
  Other Names: Routine perioperative management
  Arms: Combined Iron Supplementation Group
Procedure: Routine perioperative management — Routine perioperative management based on clinical judgment, including observation, monitoring, and standard nursing practices.
  Arms: Conventional treatment group

SUMMARY:
The goal of this clinical trial is to learn if a combined iron supplementation regimen can reduce the need for blood transfusions in adults with iron-deficiency anemia undergoing major elective cardiac surgery. The trial will also look at whether this regimen is safe and well tolerated. The main questions it aims to answer are:

Does the combined regimen lower the amount of allogeneic red blood cell transfusion needed during and after surgery?

Are there any side effects or safety concerns associated with the regimen?

Researchers will compare the combined iron supplementation (sucrose iron, erythropoietin, and vitamin C) to standard care to see if it helps reduce blood transfusions.

Participants will:

Receive either the combined regimen or standard care before surgery

Undergo major elective cardiac surgery under general anesthesia

Be monitored for blood transfusion needs and recovery up to 90 days after surgery

DETAILED DESCRIPTION:
1. Hypothesis:The combined protocol of preoperative sucrose iron, human erythropoietin, and vitamin C will demonstrate superiority in reducing perioperative allogeneic red blood cell (RBC) transfusion volume compared to standard care in patients with iron deficiency anemia undergoing major cardiac surgery with cardiopulmonary bypass.
2. Interventions 2.1.Experimental group: Patients in the experimental group will receive a combination therapy consisting of intravenous sucrose iron (200 mg), subcutaneous recombinant human erythropoietin (150 IU/kg), and intravenous vitamin C (2 g), administered once daily for three consecutive days within the week prior to surgery. All perioperative transfusion decisions will follow standardized restrictive transfusion thresholds.

   2.2.Control group: Routine perioperative management based on clinical judgment, including observation, monitoring, and standard nursing practices.
3. Primary endpoint: Total volume of allogeneic RBC transfusion (units) from surgery initiation to postoperative day 5.
4. Stratification in randomization: Stratification factors include types of surgery, preoperative baseline hemoglobin level.
5. Outcome assessors will be blinded to group allocation to reduce assessment bias.
6. Follow-up time points include: baseline upon hospital admission, the morning of surgery, postoperative day 1, postoperative day 5, at discharge, 30 ± 7 days after surgery, and 90 ± 7 days after surgery.
7. When the patient's hemoglobin concentration falls below the threshold of 70 g/L during surgery or ICU monitoring, or below 70-80 g/L in the general ward, and/or when signs of anemia or hemodynamic instability are present-including shock, severe arrhythmias, respiratory distress, heart rate >120 beats/min, systolic blood pressure (SBP) <80 mmHg, mean arterial pressure (MAP) <55-60 mmHg, or a reduction in SBP or MAP exceeding 25% from baseline-these findings may indicate significant hypovolemia and warrant consideration of transfusion intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years of age.
2. Major cardiac surgery should encompass procedures such as coronary artery bypass grafting (CABG), valve surgery, or a combination of both.
3. Iron deficiency anemia is defined as having a ferritin level below 100 μg/L or a ferritin level below 300 μg/L accompanied by a transferrin saturation below 25%. Additionally, hemoglobin levels should range between 90 and 130 g/L for men or between 90 and 120 g/L for women.
4. The American Society of Anesthesiologists (ASA) classification should fall within Grade 1-3.
5. Prior to participation, the patient or their legal representative must provide informed consent.

Exclusion Criteria:

1. Contraindications for the administration of iron sucrose, ascorbic acid, or rHuEPO.
2. Presence of a temperature exceeding 37.5 °C or the utilization of non-prophylactic antibiotics.
3. Individuals with a weight equal to or less than 50kg.
4. Individuals with a family history of haemochromatosis or thalassaemia, or those with a transferrin saturation level exceeding 50% or a documented history of iron overload.
5. Presence of other known haematological disorders such as folic acid or vitamin B12 deficiency, haemolytic anaemia, haemoglobinopathies, iron granulocytic anaemia, G6PD deficiency, etc.
6. Requirement for emergency surgical intervention.
7. Severe hepatic or renal impairment, ALT >3 times the upper limit of normal value or AST >3 times the upper limit of normal value, creatinine >1.5 times the upper limit of normal value
8. Pregnant or lactating women
9. history of blood transfusion, intravenous iron or ascorbic acid use within 12 weeks prior to surgery
10. Acute blood loss, gastrointestinal bleeding, etc. in the preoperative period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The volume of allogeneic red blood cell transfusions during the perioperative period. | From the initiation of the surgical procedure until five days post-surgery.
  The volume of allogeneic red blood cell transfusions during the perioperative period.

SECONDARY OUTCOMES:
Percentage of patients with any RBC transfusions | From the initiation of the surgical procedure until discharge. Perioperative
  The percentage of allogeneic red blood cell transfusions during the perioperative period.
Combined allogeneic transfusions (RBC, FFP( fresh frozen plasma), platelets) | From the initiation of the surgical procedure until discharge. Perioperative
  volume and Percentage
Perioperative Hb concentrations | Follow-up time points include: baseline upon hospital admission, the morning of surgery, postoperative day 1, postoperative day 5, at discharge, 30 ± 7 days after surgery, and 90 ± 7 days after surgery.
  hemoglobin
The alterations in ferritin levels and TSAT during the perioperative period. | 6.Follow-up time points include: baseline upon hospital admission, the morning of surgery, postoperative day 1, postoperative day 5, at discharge, 30 ± 7 days after surgery, and 90 ± 7 days after surgery.
  ferritin、Transferrin Saturation
The alterations in reticulocyte levels during the perioperative period. | 6.Follow-up time points include: baseline upon hospital admission, the morning of surgery, postoperative day 1, postoperative day 5, at discharge, 30 ± 7 days after surgery, and 90 ± 7 days after surgery.
  reticulocyte
The score measuring the quality of life after surgery. | From the point of randomisation until 90± 7 days following the surgical procedure.
  the results are reported using the EQ-5D-3L Effectiveness Index (EQ-5D-3L) values (5-15), where a lower EQ-5D-3L value signifies a better state of health.
Acute kidney failure | From the initiation of the surgical procedure until 7 days post-surgery.
  Acute kidney injury used to be called acute kidney failure. Acute kidney injury is most common in people who are in the hospital, mostly in people who need intensive care.
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | From the point of randomisation until 90± 7 days following the surgical procedure.
  Myocardial infarction, stroke, death
New atrial fibrillation | From the point of randomisation until 90± 7 days following the surgical procedure.
  New atrial fibrillation (AF) is defined as a new onset or a first detectable episode of AF, whether symptomatic or not
Infections | From the initiation of the surgical procedure until discharge. Perioperative
  Pneumonia, hospital acquired Deep Sternal Wound Infection
  Definition of infection: rise in inflammation markers after the initial postoperative period (acute phase reaction) and requires treatment and/ or prolongs days in hospital and/or microbiological confirmation of infection
Thrombotic and thromboembolic complications | From the initiation of the surgical procedure until discharge. Perioperative
  clinical symptoms and evidence of thrombosis/ embolism in one of the following imaging methods (ultrasound, CT-scan)
30 day and 90-day mortality | From the initiation of the surgical procedure until discharge. Perioperative
  mortality
Costs (for blood products and pharmaceutical products related to transfusion and anemia management) | From the initiation of the surgical procedure until discharge. Perioperative
  Comparison of costs for study medication versus costs for blood products and products related to transfusion
All serious adverse events | From the initiation of the surgical procedure until discharge. Perioperative
  Comparison of all serious adverse events between study intervention group and control group
Length of stay (LOS) in the hospital | Within 90± 7 days after surgery
  The time elapsed between a patient's hospital admittance and discharge
Length of stay in the intensive care unit (ICU) | Within 90± 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeroual N, Blin C, Saour M, David H, Aouinti S, Picot MC, Colson PH, Gaudard P. Restrictive Transfusion Strategy after Cardiac Surgery. Anesthesiology. 2021 Mar 1;134(3):370-380. doi: 10.1097/ALN.0000000000003682. PMID 33475735
- [Background] Fowler AJ, Ahmad T, Abbott TEF, Torrance HD, Wouters PF, De Hert S, Lobo SM, Rasmussen LS, Della Rocca G, Beattie WS, Wijeysundera DN, Pearse RM; International Surgical Outcomes Study Group. Association of preoperative anaemia with postoperative morbidity and mortality: an observational cohort study in low-, middle-, and high-income countries. Br J Anaesth. 2018 Dec;121(6):1227-1235. doi: 10.1016/j.bja.2018.08.026. Epub 2018 Oct 25. PMID 30442249
- [Background] Carson JL, Brittenham GM. How I treat anemia with red blood cell transfusion and iron. Blood. 2023 Aug 31;142(9):777-785. doi: 10.1182/blood.2022018521. PMID 36315909
- [Background] Spahn DR, Schoenrath F, Spahn GH, Seifert B, Stein P, Theusinger OM, Kaserer A, Hegemann I, Hofmann A, Maisano F, Falk V. Effect of ultra-short-term treatment of patients with iron deficiency or anaemia undergoing cardiac surgery: a prospective randomised trial. Lancet. 2019 Jun 1;393(10187):2201-2212. doi: 10.1016/S0140-6736(18)32555-8. Epub 2019 Apr 26. PMID 31036337
- [Background] Attallah N, Osman-Malik Y, Frinak S, Besarab A. Effect of intravenous ascorbic acid in hemodialysis patients with EPO-hyporesponsive anemia and hyperferritinemia. Am J Kidney Dis. 2006 Apr;47(4):644-54. doi: 10.1053/j.ajkd.2005.12.025. PMID 16564942